CLINICAL TRIAL: NCT06643052
Title: Cahnge in Management of Suspected Early Onset Neonetal Sepsis After Assimilation of Early Onset Sepsis Calculator
Status: Not yet recruiting | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Neonatologist, Hillel Yaffe Medical Center
Other Study IDs: 0121-20-HYMC-IL
Record Dates: First submitted 2024-10-14; First posted 2024-10-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Neonatal Early-onset Sepsis
Keywords: Neonatal early onset sepsis; Kaiser Permanente calculator
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before calculator: Newborn infants before assimilation of EOS calculator
  Interventions: Other: No intervention
- With calculator: Newborn infants after assimilation of EOS calculator
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Early neonatal sepsis requires rapid and efficient intervention to prevent morbidity and mortality. Management of such a case includes invasive blood examinations, elongation of maternal and neonatal length of stay, and empiric antibiotic therapy. These actions has major side effects. On 2017, Kaiser-Permanente started using a calculator that weighs the chances for early onset neonatal sepsis, and states the best investigation and follow-up regimn for the specific newborn infant. Eversince, policy of managing neonatal suspected early onset sepsis has chaged globally, including in Israel. Current knowledge regarding the local outcome since the use of the calculatir is scarce.

The goal of the study is to evaluate the change in management of suspected neonatal early onset sepsis, including its economic value, between periods before and after assimilation of the calculator in Hillel Yaffe nedica l center.

DETAILED DESCRIPTION:
Early neonatal sepsis requires rapid and efficient intervention to prevent morbidity and mortality. Management of such a case includes invasive blood examinations, elongation of maternal and neonatal length of stay, and empiric antibiotic therapy. These actions has major side effects. On 2017, Kaiser-Permanente started using a calculator that weighs the chances for early onset neonatal sepsis, and states the best investigation and follow-up regimn for the specific newborn infant. Eversince, policy of managing neonatal suspected early onset sepsis has chaged globally, including in Israel. Current knowledge regarding the local outcome since the use of the calculatir is scarce.

The goal of the study is to evaluate the change in management of suspected neonatal early onset sepsis, including its economic value, between periods before and after assimilation of the calculator in Hillel Yaffe nedical center.

ELIGIBILITY:
Inclusion Criteria:

* Newborn unfants born in Hillel Yaffe medical center
* 35 weeks of gestation or more
* Blood culture was taken

Exclusion Criteria:

* Sepsis workup for other reason
* 34 weeks of gestation or less

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants in Hillel Yaffe medical center
Sampling Method: Non-Probability Sample
Enrollment: 6300 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of negative blood cultures out of all blood cultures | during first week of life
  Total count of negative blood cultures out of all blood cultures in all patients in group
Number of positive blood cultures | during first week of life
  Total count of positive blood cultures in all patients in group

SECONDARY OUTCOMES:
Cost of treatment | during first week of life
  Total cost of Blood cultures + Blood counts + Antibiotic therpy in all patients in group

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe medical center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Did not decide yet

REFERENCES:
- [Background] Kuzniewicz MW, Puopolo KM, Fischer A, Walsh EM, Li S, Newman TB, Kipnis P, Escobar GJ. A Quantitative, Risk-Based Approach to the Management of Neonatal Early-Onset Sepsis. JAMA Pediatr. 2017 Apr 1;171(4):365-371. doi: 10.1001/jamapediatrics.2016.4678. PMID 28241253
- [Background] Hochberg A, Yehezkeli V, Nadir E, Foldi S, Feldman M. [INFECTIOUS DISEASE ASSESSMENT OF TERM INFANTS WITH RISK FACTORS - EVALUATION OF NECESSITY AND METHODS OF PREVENTION]. Harefuah. 2019 Jan;158(1):25-29. Hebrew. PMID 30663289
- [Background] Nanduri SA, Petit S, Smelser C, Apostol M, Alden NB, Harrison LH, Lynfield R, Vagnone PS, Burzlaff K, Spina NL, Dufort EM, Schaffner W, Thomas AR, Farley MM, Jain JH, Pondo T, McGee L, Beall BW, Schrag SJ. Epidemiology of Invasive Early-Onset and Late-Onset Group B Streptococcal Disease in the United States, 2006 to 2015: Multistate Laboratory and Population-Based Surveillance. JAMA Pediatr. 2019 Mar 1;173(3):224-233. doi: 10.1001/jamapediatrics.2018.4826. PMID 30640366
- [Background] Weston EJ, Pondo T, Lewis MM, Martell-Cleary P, Morin C, Jewell B, Daily P, Apostol M, Petit S, Farley M, Lynfield R, Reingold A, Hansen NI, Stoll BJ, Shane AL, Zell E, Schrag SJ. The burden of invasive early-onset neonatal sepsis in the United States, 2005-2008. Pediatr Infect Dis J. 2011 Nov;30(11):937-41. doi: 10.1097/INF.0b013e318223bad2. PMID 21654548
- [Background] Schrag SJ, Farley MM, Petit S, Reingold A, Weston EJ, Pondo T, Hudson Jain J, Lynfield R. Epidemiology of Invasive Early-Onset Neonatal Sepsis, 2005 to 2014. Pediatrics. 2016 Dec;138(6):e20162013. doi: 10.1542/peds.2016-2013. PMID 27940705